CLINICAL TRIAL: NCT05739435
Title: A Study to Evaluate the Long Term Safety and Efficacy of ESK-001 in Patients With Plaque Psoriasis
Brief Title: Open-Label Extension Study to Evaluate the Long Term Safety and Efficacy of ESK-001 in Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESK-001-007
Record Dates: First submitted 2023-02-02; First posted 2023-02-22 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ESK-001 Dose Level 1 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 2 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001

INTERVENTIONS:
Drug: ESK-001 — Oral tablet

SUMMARY:
This is a multi-center, open-label extension (OLE) study in patients with plaque psoriasis who have completed their participation in a previous plaque psoriasis study of ESK-001.

DETAILED DESCRIPTION:
This study will consist of patients who have completed their participation in a previous plaque psoriasis study of ESK-001. Each patient will be assigned to receive ESK-001 at one of two open-label dose levels. Patients have the option to remain on study until ESK-001 is commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed a prior ESK-001 study
* Men and Women must use highly effective methods of contraception for the entirety of the study

Exclusion Criteria:

* Pregnancy
* Received a prohibited concomitant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of long-term ESK-001 treatment | Approximately 3 years
  Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
To assess the long-term efficacy of ESK-001 | Approximately 3 years
  Change from baseline in Psoriasis Area and Severity Index (PASI) over time
To assess the change in quality of life (QoL) with long-term ESK-001 administration | Approximately 3 years
  Change from baseline in Dermatology Life Quality Index (DLQI) over time
To assess the pharmacokinetics (PK) of ESK-001 (ctrough) | 2 years
  Plasma concentrations and PK parameters including steady-state trough observed plasma concentration (Ctrough) for ESK-001

CONTACTS AND LOCATIONS:
Locations (38):
- United States (28):
  - Investigator Site # 1029, Birmingham, Alabama
  - Investigator Site #1001, Phoenix, Arizona
  - Investigator Site # 1023, Rogers, Arkansas
  - Investigator Site #1021, Encinitas, California
  - Investigator Site #1018, Los Angeles, California
  - Investigator Site #1007, Santa Monica, California
  - Investigator Site #1002, Sherman Oaks, California
  - Investigator site # 1030, Fort Lauderdale, Florida
  - Investigator Site #1025, Hialeah, Florida
  - Investigator site # 1028, Miami, Florida
  - Investigator Site # 1013, Tampa, Florida
  - Investigator Site #1035, Macon, Georgia
  - Investigator Site #1043, Sandy Springs, Georgia
  - Investigator Site #1005, Rolling Meadows, Illinois
  - Investigator Site # 1011, Columbus, Indiana
  - Investigator Site #1027, South Bend, Indiana
  - Investigator SIte#1036, Overland Park, Kansas
  - Investigator Site #1017, Owensboro, Kentucky
  - Investigator Site #1026, Rockville, Maryland
  - Investigator Site #1010, Clarkston, Michigan
  - Investigator Site #1031, New Brighton, Minnesota
  - Investigator Site #1033, Norman, Oklahoma
  - Investigator Site #1019, Portland, Oregon
  - Investigator Site #1022, Philadelphia, Pennsylvania
  - Investigator Site # 1012, Rapid City, South Dakota
  - Investigator Site #1015, Houston, Texas
  - Investigator Site # 1006, San Antonio, Texas
  - Investigator Site # 1041, South Jordan, Utah
- Canada (10):
  - Investigator Site #2001, Edmonton, Alberta
  - Investigator Site # 2008, Surrey, British Columbia
  - Investigator Site #2003, Winnipeg, Manitoba
  - Investigator Site #2006, London, Ontario
  - Investigator Site # 2004, Mississauga, Ontario
  - Investigator Site # 2007, North Bay, Ontario
  - Investigator Site #2005, Oakville, Ontario
  - Investigator Site #2009, Toronto, Ontario
  - Investigator Site # 2002, Waterloo, Ontario
  - Investigator Site # 2010, Québec, Quebec